## THE EFFECT OF EDUCATION GIVEN BEFORE PORT CATHETER INFUSION ON INFUSION RELATED SYMPTOMS

## KARADENİZ TECHNICAL UNIVERSITY HEALTH SCIENCES SCIENTIFIC RESEARCH ETHICS BOARD INFORMED VOLUNTEER CONSENT FORM

This form was prepared by the instructor(s) of Karadeniz Technical University, Faculty of Health Sciences, Department of Nursing, Department of Nursing Principles. The title of the study is "The Effect of Education Given Before Port Catheter Infusion on Infusion Related Symptoms" and the aim of this thesis study will be to evaluate the pain, anxiety and vital signs in patients who will start the first infusion with port catheter by giving education. Patients to be included in the study will be determined by simple randomisation method. The information provided in all interviews will be used only in this study and personal information will be kept strictly confidential. In addition, your names will definitely not be included in the research report while writing the research results. The duration of the study is 12 months. During this study, you are expected to answer the questions in the questionnaire sincerely. Below is the contact information of the researcher you can reach within the scope of the study.

| Name and Surname of the Participant (Legal representative when necessary): |
|----------------------------------------------------------------------------|
| Signature: |
| Address (if any, Phone Number): |
| Date (day/month/year):/ |

Name and Surname of the Researcher Who Made the Statements: Yekta DEMİRSOY Address: Karadeniz Technical University, Farabi Hospital Oncology Service, Ortahisar/Trabzon

Tel: 05532077477 Date (day/month/year):

Name and Surname of the Researcher Who Made the Statements: Assist. Asst. Prof. Şule Bıyık Bayram,

Address: Karadeniz Technical University, Faculty of Health Sciences, Department of Nursing,